CLINICAL TRIAL: NCT03662542
Title: A Phase 2a Randomized, Double-blind, Active-controlled, Parallel-group, Multicenter, Proof-of-concept Clinical Study to Evaluate the Efficacy and Safety of Combination Therapy With Guselkumab and Golimumab in Participants With Moderately to Severely Active Ulcerative Colitis
Brief Title: A Study of Efficacy and Safety of Combination Therapy With Guselkumab and Golimumab in Participants With Moderately to Severely Active Ulcerative Colitis
Acronym: VEGA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR108527; 2018-001510-15 (EudraCT Number); CNTO1959UCO2002 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2018-09-06; First posted 2018-09-07 (Actual); Results first posted 2023-12-12 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-11

CONDITIONS: Colitis, Ulcerative
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Combination Therapy (Experimental): Participants will receive guselkumab Dose 1 as intravenous (IV) infusion and Dose 2 as subcutaneous (SC) injection; and golimumab Dose 1 and Dose 2 as SC injection and placebo to maintain the blind.
  Interventions: Drug: Guselkumab Dose 1; Drug: Guselkumab Dose 2; Drug: Golimumab Dose 1; Drug: Golimumab Dose 2; Drug: Placebo
- Monotherapy: Guselkumab (Experimental): Participants will receive guselkumab Dose 1 as IV infusion, Dose 2 as SC injection and placebo to maintain the blind.
  Interventions: Drug: Guselkumab Dose 1; Drug: Guselkumab Dose 2; Drug: Placebo
- Monotherapy: Golimumab (Active Comparator): Participants will receive golimumab Dose 1 and Dose 2 as SC injection and placebo to maintain the blind.
  Interventions: Drug: Golimumab Dose 1; Drug: Golimumab Dose 2; Drug: Placebo

INTERVENTIONS:
Drug: Guselkumab Dose 1 — Guselkumab Dose 1 will be administered as IV infusion.
  Arms: Combination Therapy; Monotherapy: Guselkumab
Drug: Guselkumab Dose 2 — Guselkumab Dose 2 will be administered as SC injection.
  Arms: Combination Therapy; Monotherapy: Guselkumab
Drug: Golimumab Dose 1 — Golimumab Dose 1 will be administered as SC injection.
  Arms: Combination Therapy; Monotherapy: Golimumab
Drug: Golimumab Dose 2 — Golimumab Dose 2 will be administered as SC injection.
  Arms: Combination Therapy; Monotherapy: Golimumab
Drug: Placebo — Placebo will be administered.

SUMMARY:
The purpose of this study is to evaluate the clinical efficacy and safety of combination therapy with guselkumab and golimumab in participants with moderately to severely active ulcerative colitis (UC).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed clinical diagnosis of ulcerative colitis (UC) at least 3 months before screening
* Moderately to severely active UC as defined by Mayo score
* History of inadequate response to or failure to tolerate conventional therapy
* Has screening laboratory test results within the study protocol defined parameters
* A woman of childbearing potential must have a negative highly sensitive serum (beta human chorionic gonadotropin) pregnancy test result at screening and a negative urine pregnancy test result at Week 0

Exclusion Criteria:

* Has severe extensive colitis as defined in the study protocol
* Has UC limited to the rectum only or to less than (<) 20 centimeter (cm) of the colon
* Has a history of latent or active granulomatous infection, including histoplasmosis or coccidioidomycosis, before screening
* Has any known malignancy or has a history of malignancy (with the exception of basal cell carcinoma; squamous cell carcinoma in situ of the skin; or cervical carcinoma in situ that has been treated with no evidence of recurrence; or squamous cell carcinoma of the skin that has been treated with no evidence of recurrence within 5 years before screening)
* Has known allergies, hypersensitivity, or intolerance to guselkumab or golimumab or their excipients

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2018-11-20 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (82):
- United States (14):
  - Precision Research Institute, San Diego, California
  - Peak Gastroenterology Associates, Colorado Springs, Colorado
  - GCP Clinical Research, Tampa, Florida
  - Gastrointestinal Specialists of Georgia, Marietta, Georgia
  - Indiana University, Indianapolis, Indiana
  - Chevy Chase Clinical Research, Chevy Chase, Maryland
  - Woodholme Gastroenterology, Glen Burnie, Maryland
  - Sierra Clinical Research, Las Vegas, Nevada
  - The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Fargo Gastroenterology Clinic, PC, Fargo, North Dakota
  - Texas Digestive Disease Consultants, Southlake, Texas
  - Gastroenterology Associates of Tidewater, Chesapeake, Virginia
  - Virginia Mason, Seattle, Washington
  - Washington Gastroenterology, PLLC, Tacoma, Washington
- Argentina (8):
  - CEMIC (Centro de Educación Médica e Investigaciones Clínicas), Buenos Aires
  - Hospital Britanico de Buenos Aires, Buenos Aires
  - Expertia S.A, Caba
  - Centro Médico Dra. De Salvo, Caba
  - Clínica Adventista Belgrano, Ciudad de Buenos Aires
  - Fundacion de Estudios Clinicos, Rosario
  - Hospital de Alta Complejidad en Red 'El Cruce', San Juan Bautista
  - Sanatorio 9 de Julio, San Miguel de Tucumán
- Australia (7):
  - Princess Alexandra Hospital, Brisbane
  - St Vincent's Hospital - Melbourne, Fitzroy
  - Nepean Hospital, Kingswood
  - Royal Adelaide Hospital, North Terrace
  - Macquarie University Hospital, NSW
  - Royal Melbourne Hospital, Parkville
  - Mater Hospital Brisbane (Inflammatory Bowel Diseases), South Brisbane
- Brazil (10):
  - Hospital Das Clinicas Da Ufmg, Belo Horizonte
  - Universidade Estadual Paulista 'Julio De Mesquita Filho', Botucatu
  - Inst Goiano Gastroenterologia e Endoscopia Digest Ltda - Clinica de Gastro, Goiânia
  - Hospital das Clinicas de Porto Alegre, Porto Alegre
  - Hospital das Clínicas da Faculdade de Medicina de RPUSP - HCRP, Ribeirão Preto
  - Universidade Federal do Rio de Janeiro - Faculdade de Medicina, Rio de Janeiro
  - Instituto Brasil de Pesquisa Clinica, Rio de Janeiro
  - Fundacao do ABC - Centro Universitario FMABC, Santo André
  - Kaiser Hospta, São José do Rio Preto
  - Eurolatino Pesquisas Medicas Ltda, Uberlândia
- Germany (4):
  - Charite Berlin, Berlin
  - Universitatsklinikum Frankfurt/ Medizinische Klinik 1, Frankfurt
  - Universitätsklinikum Jena, Jena
  - Universitaetsklinikum Ulm, Ulm
- Mexico (5):
  - Clínica Saluz, Boca del Rio
  - Clinicos Asociados BOCM, SC, Mexico City
  - Centro Regiomontano de Estudios Clínicos Roma S.C., Monterrey
  - Capital Humano para la Investigacion clinica, Querétaro
  - Centro Medico Zambrano Hellion, San Pedro Garza García
- Poland (8):
  - Synexus Polska Sp. z o.o. Oddzial w Gdansku, Gdansk
  - Pratia MCM Krakow, Krakow
  - Endoskopia Sp. z o.o. z siedzibą w Sopocie, Sopot
  - Centrum Zdrowia MDM, Warsaw
  - WIP Warsaw IBD Point Profesor Kierkus, Warsaw
  - Centralny Szpital Kliniczny MSWiA w Warszawie, Warsaw
  - Niepubliczny Zakład Opieki Zdrowotnej Vivamed Jadwiga Miecz, Warsaw
  - Melita Medical Sp. z o.o., Wroclaw
- Russia (14):
  - Kazan State Medical University, Kazan'
  - City Clinical Hospital # 24, Moscow
  - Medical Center SibNovoMed LLC, Novosibirsk
  - Rostov State Medical University, Rostov-on-Don
  - International Medical Centre SOGAZ, Saint Petersburg
  - Elizavetinskaya hospital, Saint Petersburg
  - Eco-safety Ltd, Saint Petersburg
  - City Clinical Hospital #31, Saint Petersburg
  - Medical University Reaviz, Samara
  - Tver Regional Clinical Hospital, Tver'
  - GBUZ Respublican Clinical Hospital n.a. GG Kuvatova, Ufa
  - City Clinical Hospital #2, Yaroslavl
  - Regional Clinical Hospital, Yaroslavl
  - Medical Association 'New Hospital', Yekaterinburg
- Ukraine (12):
  - Communal Nonprofit Enterprise 'City Clinical Hospital # 2 N.A. Prof. O.O. Shalimov', Kharkiv
  - SI 'L.T. Maloyi National Institute of Therapy of National Academy of Medical Sciences of Ukraine, Kharkiv
  - Municipal Institution 'Kherson City Clinical Hospital n.a. Y.Y.Karabelesh', Kherson
  - Kyiv City Clinical Hospital #18, Kyiv
  - Medical Center 'Ok Clinic' of LLC 'International Institute of Clinical Studies', Kyiv
  - Lviv Clinical Hospital on Railway Transport of Affiliate Healthcare center of JSC Ukrainian Railway, Lviv
  - Communal Nonprofit Enterprise of Lviv Regional Council 'Lviv Regional Clinical Hospital', Lviv
  - Municipal Non-profit Enterprise 'Odesa Regional Clinical Hospital' Odesa Regional Council, Odesa
  - Sumy State University, Sumy Regional Clinical Hospital, Sumy
  - Municipal institution of Tepnopil Regional Council 'Ternopil University Hospital', Ternopil
  - Medical Center Ltd 'Health Clinic', Department Of General Therapy, Vinnytsia
  - Vinnitsia Regional Clinical Hospital n.a. M. I. Pyrogov, Vinnytsia

REFERENCES:
- [Derived] Shao J, Vetter M, Vermeulen A, Feagan BG, Sands BE, Panes J, Xu Z. Combination Therapy With Guselkumab and Golimumab in Patients With Moderately to Severely Active Ulcerative Colitis: Pharmacokinetics, Immunogenicity and Drug-Drug Interactions. Clin Pharmacol Ther. 2024 Jun;115(6):1418-1427. doi: 10.1002/cpt.3235. Epub 2024 Mar 15. PMID 38488354
- [Derived] Feagan BG, Sands BE, Sandborn WJ, Germinaro M, Vetter M, Shao J, Sheng S, Johanns J, Panes J; VEGA Study Group. Guselkumab plus golimumab combination therapy versus guselkumab or golimumab monotherapy in patients with ulcerative colitis (VEGA): a randomised, double-blind, controlled, phase 2, proof-of-concept trial. Lancet Gastroenterol Hepatol. 2023 Apr;8(4):307-320. doi: 10.1016/S2468-1253(22)00427-7. Epub 2023 Feb 1. PMID 36738762

RESULTS

PARTICIPANT FLOW:
Groups:
- Combination Phase: Golimumab Monotherapy: Participants received golimumab 200 milligrams (mg) as subcutaneous (SC) injection at Week 0, followed by golimumab 100 mg as SC injection at Weeks 2, 6 and 10. Participants received placebo as intravenous (IV) infusion at Weeks 0, 4 and 8 to maintain the blind. Participants were then assessed for efficacy at Week 10 and Week 12.
- Combination Phase: Guselkumab Monotherapy: Participants received guselkumab 200 mg as IV infusion at Weeks 0, 4 and 8. Participants received placebo as SC injection at Weeks 0, 2, 6 and 10 to maintain the blind. Participants were then assessed for efficacy at Week 10 and Week 12.
- Combination Phase: Combination Therapy: Participants received guselkumab 200 mg as IV infusion at Weeks 0, 4, and 8. Participants received golimumab 200 mg as SC injection at Week 0, followed by golimumab 100 mg as SC injection at Weeks 2, 6 and 10. Participants were then assessed for efficacy at Week 10 and Week 12.
- Monotherapy Phase: Golimumab Monotherapy: Participants received golimumab 100 mg as SC injection at Weeks 14, 18, 22, 26, 30 and 34, and placebo as SC injection at Weeks 16, 24, and 32 to maintain the blind. Participants were then assessed for efficacy at Week 38.
- Monotherapy Phase: Guselkumab Monotherapy: Participants received guselkumab 100 mg as SC injection at Weeks 16, 24, and 32, and placebo as SC injection at Weeks 14, 18, 22, 26, 30, and 34 to maintain the blind. Participants were then assessed for efficacy at Week 38.
- Monotherapy Phase: Combination Therapy: Participants received guselkumab 100 mg as SC injection at Weeks 16, 24 and 32, and placebo as SC injection at Weeks 14, 18, 22, 26, 30, and 34 to maintain the blind. Participants were then assessed for efficacy at Week 38.
- Safety Follow-up: Golimumab Monotherapy: Participants were followed up for safety from Week 38 to Week 50 (end of study [EOS]) and did not receive any additional medication in the safety follow-up phase.
- Safety Follow-up: Guselkumab Monotherapy; Safety Follow-up: Combination Therapy: Participants were followed up for safety from Week 38 to Week 50 (EOS) and did not receive any additional medication in the safety follow-up phase.
Period: Combination Phase ( Week 0- Week 12)
Arm/Group | Combination Phase: Golimumab Monotherapy | Combination Phase: Guselkumab Monotherapy | Combination Phase: Combination Therapy | Monotherapy Phase: Golimumab Monotherapy | Monotherapy Phase: Guselkumab Monotherapy | Monotherapy Phase: Combination Therapy | Safety Follow-up: Golimumab Monotherapy | Safety Follow-up: Guselkumab Monotherapy | Safety Follow-up: Combination Therapy
Started | 72 | 71 | 71 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 67 | 70 | 71 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 5 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — COVID-19 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Monotherapy Phase (Week 12-Week 38)
Arm/Group | Combination Phase: Golimumab Monotherapy | Combination Phase: Guselkumab Monotherapy | Combination Phase: Combination Therapy | Monotherapy Phase: Golimumab Monotherapy | Monotherapy Phase: Guselkumab Monotherapy | Monotherapy Phase: Combination Therapy | Safety Follow-up: Golimumab Monotherapy | Safety Follow-up: Guselkumab Monotherapy | Safety Follow-up: Combination Therapy
Started | 0 | 0 | 0 | 67 | 70 | 71 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 62 | 67 | 65 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 5 | 3 | 6 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 4 | 1 | 1 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Period: Safety Follow-up (Week 38- Week 50)
Arm/Group | Combination Phase: Golimumab Monotherapy | Combination Phase: Guselkumab Monotherapy | Combination Phase: Combination Therapy | Monotherapy Phase: Golimumab Monotherapy | Monotherapy Phase: Guselkumab Monotherapy | Monotherapy Phase: Combination Therapy | Safety Follow-up: Golimumab Monotherapy | Safety Follow-up: Guselkumab Monotherapy | Safety Follow-up: Combination Therapy
Started | 0 | 0 | 0 | 0 | 0 | 0 | 58 (Participants could be followed up even if they did not complete treatment.) | 65 (Participants could be followed up even if they did not complete treatment.) | 60 (Participants could be followed up even if they did not complete treatment.)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 55 | 58 | 55
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 7 | 5
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 6 | 2

BASELINE CHARACTERISTICS:
Groups:
- Golimumab Monotherapy: Participants received golimumab 200 milligrams (mg) as subcutaneous (SC) injection at Week 0 followed by golimumab 100 mg as SC injection at Weeks 2, 6, 10, 14, 18, 22, 26, 30 and 34. Participants received placebo as intravenous (IV) infusion as Weeks 0, 4, 8 and as SC injection at Weeks 16, 24, 32 to maintain the blind. Participants were then followed up for safety from Week 38 to Week 50 (end of study [EOS]).
- Guselkumab Monotherapy: Participants received guselkumab 200 mg as IV infusion at Weeks 0, 4 and 8 followed by guselkumab 100 mg as SC injection at Weeks 16, 24 and 32. Participants received placebo as SC injection at Weeks 0, 2, 6, 10, 14, 18, 22, 26, 30, and 34 to maintain the blind. Participants were then followed up for safety from Week 38 to Week 50 (EOS).
- Combination Therapy: Participants received guselkumab 200 mg as IV infusion followed by golimumab 200 mg as SC injection at Weeks 0. Participants received guselkumab 200 mg as IV infusion at Weeks 4 and 8, golimumab 100 mg as SC injection at Weeks 2, 6 and 10 and placebo as SC injection at Weeks 14, 18, 22, 26, 30, and 34 to maintain the blind. Participants were then followed up for safety from Week 38 to Week 50 (EOS).
- Total: Total of all reporting groups
Arm/Group | Golimumab Monotherapy | Guselkumab Monotherapy | Combination Therapy | Total
Number analyzed (Participants) | 72 | 71 | 71 | 214
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 72 | 70 | 71 | 213
  >=65 years | 0 | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.1 (10.47) | 39.1 (13.67) | 37.8 (11.69) | 38.4 (11.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 31 | 37 | 98
  Male | 42 | 40 | 34 | 116
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 6 | 5 | 15
  Not Hispanic or Latino | 68 | 65 | 66 | 199
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 0 | 2
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 0 | 1 | 4
  White | 67 | 71 | 70 | 208
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  ARGENTINA | 0 | 1 | 3 | 4
  AUSTRALIA | 2 | 1 | 1 | 4
  BRAZIL | 2 | 3 | 4 | 9
  GERMANY | 0 | 1 | 1 | 2
  MEXICO | 2 | 2 | 0 | 4
  POLAND | 15 | 11 | 14 | 40
  RUSSIAN FEDERATION | 19 | 22 | 30 | 71
  UKRAINE | 27 | 25 | 16 | 68
  UNITED STATES | 5 | 5 | 2 | 12

OUTCOME MEASURES:

1. Primary Outcome: Combination Phase: Percentage of Participants Who Achieved Clinical Response at Week 12
Description: Clinical response was defined as a decrease from baseline in the Mayo score greater than or equal to (>=) 30 percent (%) and >=3 points with either a decrease from baseline in the rectal bleeding subscore (RBS) >=1 or a RBS of 0 or 1. The Mayo score was calculated as the sum of 4 subscores (stool frequency, rectal bleeding, physician's global assessment, and endoscopy findings - each with score range of 0 (normal activity) to 3 (severe activity) and a total score range of 0 to 12 points. A score of 3 to 5 points indicates mildly active disease, a score of 6 to 10 points indicates moderately active disease, and a score of 11 to 12 points indicates severely active disease. Higher scores indicate more severity. This outcome measure was analyzed for combination phase only as preplanned in the protocol.
Time Frame: Week 12
Population: Efficacy analyses were based on the full analysis set (FAS), which included all randomized participants who received at least 1 (partial or complete) dose of study intervention.
Measure: Number; unit: Percentage of participants
Arm/Group | Combination Phase: Golimumab Monotherapy | Combination Phase: Guselkumab Monotherapy | Combination Phase: Combination Therapy
Number analyzed (Participants) | 72 | 71 | 71
Percentage of participants | 61.1 | 74.6 | 83.1

2. Secondary Outcome: Combination Phase: Percentage of Participants Who Achieved Clinical Remission at Week 12
Description: Clinical remission was defined as the Mayo score less than or equal to (<=) 2 with no individual subscore greater than (>) 1. The Mayo score was calculated as the sum of 4 subscores (stool frequency, rectal bleeding, physician's global assessment, and endoscopy findings) each with score range of 0 (normal activity) to 3 (severe activity) and a total score range of 0 to 12 points. A score of 3 to 5 points indicates mildly active disease, a score of 6 to 10 points indicates moderately active disease, and a score of 11 to 12 points indicates severely active disease. Higher scores indicate more severity. This outcome measure was analyzed for combination phase only as preplanned in the protocol.
Time Frame: Week 12
Population: Efficacy analyses were based on the FAS, which included all randomized participants who received at least 1 (partial or complete) dose of study intervention.
Measure: Number; unit: Percentage of participants
Arm/Group | Combination Phase: Golimumab Monotherapy | Combination Phase: Guselkumab Monotherapy | Combination Phase: Combination Therapy
Number analyzed (Participants) | 72 | 71 | 71
Percentage of participants | 22.2 | 21.1 | 36.6

ADVERSE EVENTS:
Time Frame: Up to Week 50
Description: The safety analysis set included all randomized participants who received at least 1 (partial or complete) dose of study intervention.
Arm/Group | Combination Phase: Golimumab Monotherapy | Combination Phase: Guselkumab Monotherapy | Combination Phase: Combination Therapy | Monotherapy Phase: Golimumab Monotherapy | Monotherapy Phase: Guselkumab Monotherapy | Monotherapy Phase: Combination Therapy | Safety Follow-up: Golimumab Monotherapy | Safety Follow-up: Guselkumab Monotherapy | Safety Follow-up: Combination Therapy
All-Cause Mortality (participants affected / at risk) | 0/72 | 0/71 | 0/71 | 0/67 | 0/70 | 1/71 | 0/58 | 1/65 | 0/60
Serious Adverse Events (participants affected / at risk) | 1/72 | 2/71 | 1/71 | 3/67 | 1/70 | 3/71 | 0/58 | 2/65 | 0/60
Other Adverse Events (participants affected / at risk) | 19/72 | 16/71 | 14/71 | 12/67 | 16/70 | 14/71 | 3/58 | 2/65 | 0/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Combination Phase: Golimumab Monotherapy (N=72) | Combination Phase: Guselkumab Monotherapy (N=71) | Combination Phase: Combination Therapy (N=71) | Monotherapy Phase: Golimumab Monotherapy (N=67) | Monotherapy Phase: Guselkumab Monotherapy (N=70) | Monotherapy Phase: Combination Therapy (N=71) | Safety Follow-up: Golimumab Monotherapy (N=58) | Safety Follow-up: Guselkumab Monotherapy (N=65) | Safety Follow-up: Combination Therapy (N=60)
Atrial Fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colitis Ulcerative (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chronic Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Covid-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Covid-19 Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tuberculosis of Intrathoracic Lymph Nodes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Adenocarcinoma of Colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Combination Phase: Golimumab Monotherapy (N=72) | Combination Phase: Guselkumab Monotherapy (N=71) | Combination Phase: Combination Therapy (N=71) | Monotherapy Phase: Golimumab Monotherapy (N=67) | Monotherapy Phase: Guselkumab Monotherapy (N=70) | Monotherapy Phase: Combination Therapy (N=71) | Safety Follow-up: Golimumab Monotherapy (N=58) | Safety Follow-up: Guselkumab Monotherapy (N=65) | Safety Follow-up: Combination Therapy (N=60)
Anaemia (Blood and lymphatic system disorders) | 5 | 6 | 4 | 2 | 6 | 0 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 4 | 2 | 1 | 2 | 2 | 0 | 0 | 0
Colitis Ulcerative (Gastrointestinal disorders) | 8 | 1 | 4 | 5 | 4 | 6 | 3 | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 4 | 5 | 1 | 2 | 2 | 6 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 3 | 4 | 2 | 5 | 3 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2019-03-07): https://cdn.clinicaltrials.gov/large-docs/42/NCT03662542/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-24): https://cdn.clinicaltrials.gov/large-docs/42/NCT03662542/SAP_001.pdf